CLINICAL TRIAL: NCT01382966
Title: The Association of Serum Sclerostin Levels,Echocardiographic Parameters, Arteriovenous Fistula Thrombosis and Carpal Tunnel Syndrome in Maintenance Hemodialysis Patients
Brief Title: Serum Sclerostin Levels, Cardiovascular Parameters and Carpal Tunnel Syndrome in Maintenance Hemodialysis Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: RFM Renal Treatment Services (Other)
Responsible Party: RFM RENAL TEDAVİ HİZMETLERİ, RFM RENAL TEDAVİ HİZMETLERİ
Other Study IDs: RFM RENAL
Record Dates: First submitted 2011-06-21; First posted 2011-06-27 (Estimated); Last update posted 2011-06-28 (Estimated); Status verified 2011-06

CONDITIONS: Chronic Kidney Disease; Renal Osteodystrophy; Left Ventricular Hypertrophy
Keywords: sclerostin; arteriovenous fistula thrombosis; carpal tunnel syndrome; echocardiography
MeSH Terms: conditions — Renal Insufficiency, Chronic; Chronic Kidney Disease-Mineral and Bone Disorder; Hypertrophy, Left Ventricular; Sclerosteosis; Carpal Tunnel Syndrome

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Single group: Maintenance hemodialysis patients of minimal 6 months of hemodialysis duration; free of malignancy, infection and autoimmune disease; age over 18 years

SUMMARY:
Sclerostin, the product of the SOST gene, located on chromosome 17, locus q11.2 in humans, was originally believed to be a non-classical Bone morphogenetic protein (BMP) antagonist.Sclerostin was recently identified as a component of parathyroid hormone (PTH) signal transduction.

Chronic kidney disease (CKD) is associated with abnormalities in bone and mineral metabolism.New advances in the pathogenesis of renal osteodystrophy (ROD) change the perspective from which many of its features and treatment are viewed. Calcium, phosphate, parathyroid hormone (PTH), and vitamin D have been shown to be important determinants of survival associated with kidney diseases. Now ROD dependent and independent of these factors is linked to survival more than just skeletal frailty.Furthermore, ROD is shown to be an underappreciated factor in the level of the serum phosphorus in CKD. The discovery and the elucidation of the mechanism of hyperphosphatemia as a cardiovascular risk in CKD change the view of ROD.

Emerging current data suggests a promising role for serum measurements of sclerostin in addition to iPTH in the diagnosis of high bone turnover in chronic kidney disease-5D patients (dialysis patients).

Because of the close relationship between ROD and cardiovascular disease, the aim of this study is to investigate the association between sclerostin, arteriovenous fistula thrombosis, echocardiography and carpal tunnel syndrome in maintenance hemodialysis patients.

DETAILED DESCRIPTION:
Sclerostin, the product of the SOST gene, located on chromosome 17, locus q11.2 in humans, was originally believed to be a non-classical Bone morphogenetic protein (BMP) antagonist.More recently Sclerostin has been identified as binding to LRP5/6 receptors and inhibiting the Wnt signalling pathway .Wnt activation under these circumstances is antagonistic to bone formation. Although the underlying mechanisms are unclear, it is believed that the antagonism of BMP-induced bone formation by sclerostin is mediated by Wnt signalling, but not BMP signalling pathways.

Sclerostin is produced by the osteocyte and has catabolic effects on bone formation. This protein, with a length of 113 residues, has a dssp secondary structure that is 28% beta sheet (6 strands; 32 residues. Sclerostin has an inhibitory effect on the lifetime of the osteoblast. Sclerostin production by osteocytes is inhibited by parathyroid hormone, mechanical loading and cytokines including oncostatin M, cardiotrophin-1 and leukemia inhibitory factor. Sclerostin production is increased by calcitonin. Thus, osteoblast activity is self regulated by a negative feedback system.Sclerostin was recently identified as a component of parathyroid hormone (PTH) signal transduction.

Chronic kidney disease (CKD) is associated with abnormalities in bone and mineral metabolism.Renal osteodystrophy (ROD) is one of the three components of chronic kidney disease-mineral and bone disorder (CKD-MBD. Patients with CKD may develop various types of bone disease, spanning the spectrum of extreme situations such as severe osteitis fibrosa, osteomalacia, mixed osteopathy, and adynamic bone disease. In addition, patients may have osteoporosis, which increases the risk for fractures, both in advanced and in less severe CKD stages (2- 4),which, in turn, result in excess mortality New advances in the pathogenesis of renal osteodystrophy (ROD) change the perspective from which many of its features and treatment are viewed. Calcium, phosphate, parathyroid hormone (PTH), and vitamin D have been shown to be important determinants of survival associated with kidney diseases. Now ROD dependent and independent of these factors is linked to survival more than just skeletal frailty.Furthermore, ROD is shown to be an underappreciated factor in the level of the serum phosphorus in CKD. The discovery and the elucidation of the mechanism of hyperphosphatemia as a cardiovascular risk in CKD change the view of ROD. Emerging current data suggests a promising role for serum measurements of sclerostin in addition to iPTH in the diagnosis of high bone turnover in chronic kidney disease-5D patients (dialysis patients).

The demonstration that the level of serum sclerostin,which is directly produced by osteocytes, is a good predictor for bone formation in patients with CKD may be of clinical interest.Because of the close relationship between ROD and cardiovascular disease, the aim of this study is to investigate the association between sclerostin, arteriovenous fistula thrombosis, echocardiography and carpal tunnel syndrome in maintenance hemodialysis patients.

ELIGIBILITY:
Inclusion Criteria:

* Maintenance hemodialysis patients (minimum 6 months of duration)
* Willingness
* Age > 18 years

Exclusion Criteria:

* Infection
* Malignancy
* Autoimmune disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Maintenance hemodialysis patients (minimum 6 months of duration) No infection, malignancy and autoimmune disease Age> 18 years
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2011-07; Primary Completion 2011-09 (Estimated); Study Completion 2011-10 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with left ventricular hypertrophy or left ventricular dysfunction according to tertiles of the serum sclerostin levels | 3 months

SECONDARY OUTCOMES:
Number of Participants with arteriovenous fistula thrombosis | 3 months
Number of Participants with carpal tunnel syndrome according to tertiles of the serum sclerostin levels | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: ALPER KIRKPANTUR, MD, Principal Investigator — RFM Renal Treatment Services
Locations (1):
- Rfm Renal Tedavi Merkezi, Ankara, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] Drueke TB, Lafage-Proust MH. Sclerostin: just one more player in renal bone disease? Clin J Am Soc Nephrol. 2011 Apr;6(4):700-3. doi: 10.2215/CJN.01370211. Epub 2011 Mar 24. No abstract available. PMID 21441122
- [Background] Cejka D, Herberth J, Branscum AJ, Fardo DW, Monier-Faugere MC, Diarra D, Haas M, Malluche HH. Sclerostin and Dickkopf-1 in renal osteodystrophy. Clin J Am Soc Nephrol. 2011 Apr;6(4):877-82. doi: 10.2215/CJN.06550810. Epub 2010 Dec 16. PMID 21164019
- [Background] Cejka D, Jager-Lansky A, Kieweg H, Weber M, Bieglmayer C, Haider DG, Diarra D, Patsch JM, Kainberger F, Bohle B, Haas M. Sclerostin serum levels correlate positively with bone mineral density and microarchitecture in haemodialysis patients. Nephrol Dial Transplant. 2012 Jan;27(1):226-30. doi: 10.1093/ndt/gfr270. Epub 2011 May 25. PMID 21613383
- [Derived] Kirkpantur A, Balci M, Turkvatan A, Afsar B. Serum sclerostin levels, arteriovenous fistula calcification and 2-years all-cause mortality in prevalent hemodialysis patients. Nefrologia. 2016;36(1):24-32. doi: 10.1016/j.nefro.2015.07.006. Epub 2015 Nov 3. PMID 26546060